CLINICAL TRIAL: NCT01837147
Title: Using Technology to Promote Activity in Women at Elevated Breast Cancer Risk
Brief Title: Using Technology to Improve Physical Activity Levels Among Postmenopausal Women (The Active & Aware Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R03CA168450-01 (NIH)
Record Dates: First submitted 2013-04-06; First posted 2013-04-23 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: primary prevention; sedentary; overweight; obesity; breast cancer; post-menopausal; women
MeSH Terms: conditions — Breast Neoplasms; Sedentary Behavior; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based Tracking Group (Experimental): Technology-Based Physical Activity Promotion
  Interventions: Behavioral: Technology-Based Physical Activity Promotion
- Pedometer Group (Active Comparator): Participants assigned to this group will receive a pedometer.
  Interventions: Behavioral: Pedometer Intervention

INTERVENTIONS:
Behavioral: Technology-Based Physical Activity Promotion — Participants assigned to this group will use a web-integrated physical activity monitor, and accompanying website, to improve their physical activity levels.
  Arms: Web-based Tracking Group
Behavioral: Pedometer Intervention — Participants assigned to this group will receive a pedometer and be trained in its use.
  Arms: Pedometer Group

SUMMARY:
Women who are overweight or do not exercise are at higher risk for breast cancer after menopause. This study will test a new electronic device that measures the body's movement and works alongside a website to help women increase their physical activity level. If effective, this system could be tested in larger studies aiming to reduce breast cancer risk by reducing or preventing obesity.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Postmenopausal
* BMI >= 25.0 kg/m2
* Physically inactive
* Internet user with regular access to high-speed internet
* Willing and able to complete study requirements

Exclusion Criteria:

* History of invasive breast cancer
* Medical contraindication to exercise
* Medical problem or other issue that would interfere with intervention
* Current participation in another physical activity study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in objectively-measured physical activity | Baseline to 16 weeks
  Assessed using ActiGraph.

SECONDARY OUTCOMES:
Self-reported physical activity | Baseline to 16 weeks
  Assessed using questionnaires.
Body weight (kg) | Baseline to 16 weeks
  Measured in clinic.
Uptake of technology-based intervention components | During 16-week intervention
  To be assessed via data downloaded from the website used in this study.
Quality of life | Baseline to 16 weeks
  To be assessed via self-report questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Cadmus-Bertram, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

REFERENCES:
- [Derived] Cadmus-Bertram L, Marcus BH, Patterson RE, Parker BA, Morey BL. Use of the Fitbit to Measure Adherence to a Physical Activity Intervention Among Overweight or Obese, Postmenopausal Women: Self-Monitoring Trajectory During 16 Weeks. JMIR Mhealth Uhealth. 2015 Nov 19;3(4):e96. doi: 10.2196/mhealth.4229. PMID 26586418
- [Derived] Cadmus-Bertram LA, Marcus BH, Patterson RE, Parker BA, Morey BL. Randomized Trial of a Fitbit-Based Physical Activity Intervention for Women. Am J Prev Med. 2015 Sep;49(3):414-8. doi: 10.1016/j.amepre.2015.01.020. Epub 2015 Jun 10. PMID 26071863